CLINICAL TRIAL: NCT06934772
Title: Comparison of the Analgesic Efficacy of Subcostal Transversus Abdominis Plane and Modified Thoracoabdominal Nerves Block Through Perichondrial Approach (M-TAPA) Blocks in Laparoscopic Sleeve Gastrectomy Surgery
Brief Title: Comparison of the Analgesic Efficacy of Subcostal TAP and M-TAPA Blocks in Laparoscopic Sleeve Gastrectomy Surgery
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Munevver Kayhan, Lecturer doctor, Istanbul University - Cerrahpasa
Other Study IDs: HEA-AAR-MK-04
Record Dates: First submitted 2025-04-05; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Plane Block; Regional Anaesthesia; Transversus Abdominis Plane (TAP) Block; Bariatric Surgery
Keywords: perioperative pain management; M-TAPA block; peripheral plane block; pain management, bariatric surgery
MeSH Terms: conditions — Bites and Stings; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- M-TAPA Group: Patients who were applied M-TAPA the inclusion criteria will be included in the study, and data will be retrospectively reviewed. Intraoperative hemodynamic data, surgical duration, and total opioid consumption will be collected from anesthesia records. Postoperative analgesic use and pain scores will be assessed from nurse documentation and medical records. Patients with incomplete data or pre-existing chronic pain conditions will be excluded.
  Interventions: Other: M-TAPA
- Subcostal TAP Group: Patients who were applied M-TAPA the inclusion criteria will be included in the study, and data will be retrospectively reviewed. Intraoperative hemodynamic data, surgical duration, and total opioid consumption will be collected from anesthesia records. Postoperative analgesic use and pain scores will be assessed from nurse documentation and medical records. Patients with incomplete data or pre-existing chronic pain conditions will be excluded.
  Interventions: Other: Subcostal TAP

INTERVENTIONS:
Other: M-TAPA — this study will be compare the analgesic efficacy of bilateral subcostal transversus abdominis plane (TAP) and modified thoracoabdominal (M-TAPA) blocks in reducing intraoperative opioid consumption and postoperative analgesic needs in patients undergoing laparoscopic sleeve gastrectomy (LSG).
  Groups: M-TAPA Group
Other: Subcostal TAP — this study will be compare the analgesic efficacy of bilateral subcostal transversus abdominis plane (TAP) and modified thoracoabdominal (M-TAPA) blocks in reducing intraoperative opioid consumption and postoperative analgesic needs in patients undergoing laparoscopic sleeve gastrectomy (LSG).
  Groups: Subcostal TAP Group

SUMMARY:
Objective The aim of this study is to compare the analgesic efficacy of bilateral subcostal transversus abdominis plane (TAP) and modified thoracoabdominal (M-TAPA) blocks in reducing intraoperative opioid consumption and postoperative analgesic needs in patients undergoing laparoscopic sleeve gastrectomy (LSG). This will be a retrospective study conducted at Haseki Training and Research Hospital between January and November 2024. The study will include patients with a Body mass index (BMI) greater than 35 kg/m², aged between 18 and 65, who are scheduled to undergo LSG surgery. Patients will receive either a subcostal TAP or M-TAPA block before surgery. Data will be collected from patient records, including intraoperative opioid usage, postoperative analgesic consumption, and pain scores (NRS) assessed at rest and during activity in the first 24 hours. Secondary outcomes will include mobilization times and incidence of postoperative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
Objective The aim of this study is to compare the analgesic efficacy of bilateral subcostal transversus abdominis plane (TAP) and modified thoracoabdominal (M-TAPA) blocks in reducing intraoperative opioid consumption and postoperative analgesic needs in patients undergoing laparoscopic sleeve gastrectomy (LSG).

Study Design This will be a retrospective study conducted at Haseki Training and Research Hospital between January and November 2024. The study will include patients with a BMI greater than 35 kg/m², aged between 18 and 65, who are scheduled to undergo LSG surgery. Patients will receive either a subcostal TAP or M-TAPA block before surgery. Data will be collected from patient records, including intraoperative opioid usage, postoperative analgesic consumption, and pain scores (NRS) assessed at rest and during activity in the first 24 hours. Secondary outcomes will include mobilization times and incidence of postoperative nausea and vomiting (PONV).

Study Procedures Patients who meet the inclusion criteria will be included in the study, and data will be retrospectively reviewed. Intraoperative hemodynamic data, surgical duration, and total opioid consumption will be collected from anesthesia records. Postoperative analgesic use and pain scores will be assessed from nurse documentation and medical records. Patients with incomplete data or pre-existing chronic pain conditions will be excluded.

Outcome Measures

* Primary Outcome: Comparison of the analgesic efficacy of M-TAPA and subcostal TAP blocks during intraoperative and postoperative periods (first 24 hours).
* Secondary Outcomes: Resting and active NRS pain scores, mobilization times, incidence of nausea and vomiting, and complications related to the block procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients with a BMI greater than 35 kg/m²,
* aged between 18 and 65, who are scheduled to undergo LSG surgery.
* Patients will receive either a subcostal TAP or M-TAPA block before surgery. Exclusion Criteria:
* patients with incomplete data
* patients with chronic pain
* patients with preoperative opioid use
* patients with preoperative alcohol/substance use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a body mass index (BMI) >35 kg/m², Charlson comorbidity index <4, who had received either a subcostal TAP or M-TAPA block after induction but prior to laparoscopic sleeve gastrectomy surgery were included.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Analgesic Efficacy | Intraoperative periods, postoperative first 24 hours.
  Comparison of the analgesic efficacy of M-TAPA and subcostal TAP blocks during intraoperative and postoperative periods.The visual pain score includes values between 0 and 10. o means no pain, 5 means moderate pain, and 10 means severe pain. In the postoperative period, the pain levels of the patients will be compared by looking at this visual pain value. In the intraoperative period, the amount of analgesic consumption (total consumption of remifentanil mcg) will be evaluated.

SECONDARY OUTCOMES:
Other conditions associated with the block | postoperative 24 hours
  Resting and active NRS pain scores, mobilization times, nausea and vomiting frequency and complications related to block procedures. Visual pain scores of patients when they first start moving postoperatively will be examined. 0 is evaluated as no pain, 5 as moderate pain, 10 as very severe pain. The time they first started mobilizing will be determined according to the postoperative hour. It will be recorded as whether nausea and vomiting occurred or not. If there were other complications (e.g. bleeding at the block site, hematoma, shortness of breath, pneumothorax), all this information will be determined from the patient files.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turunc E, Dost B, Sarikaya Ozel E, Kaya C, Ustun YB, Bilgin S, Ozbalci GS, Koksal E. Bilateral Ultrasound-Guided External Oblique Intercostal Block Vs. Modified Thoracoabdominal Nerve Block Through Perichondrial Approach for Postoperative Analgesia in Patients Undergoing Laparoscopic Sleeve Gastrectomy Surgery: A Randomized Controlled Study. Obes Surg. 2024 Oct;34(10):3726-3734. doi: 10.1007/s11695-024-07454-4. Epub 2024 Sep 11. PMID 39259439